CLINICAL TRIAL: NCT03842007
Title: Understanding Mechanisms of Normal and Disordered Defecation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Adil Bharucha, MBBS, MD, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-010327; R01DK078924 (NIH)
Record Dates: First submitted 2019-01-10; First posted 2019-02-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Individuals (Active Comparator): Sixty healthy individuals (20 men and 40 women) will undergo an anorectal study which comprises of a rectal barostat study followed by fecoflowmetry
  Interventions: Diagnostic Test: Rectal Barostat Study; Diagnostic Test: Fecoflowmetry
- Constipated Individuals (Active Comparator): 60 constipated individuals (20 men and 40 women) will undergo an anorectal study which comprises of a rectal barostat study followed by fecoflowmetry
  Interventions: Diagnostic Test: Rectal Barostat Study; Diagnostic Test: Fecoflowmetry

INTERVENTIONS:
Diagnostic Test: Rectal Barostat Study — Contractions will be recorded with a balloon inserted into the rectum and inflated
Diagnostic Test: Fecoflowmetry — Rectum will be filled with a small amount of paste.Two thin catheters will be inserted into the anus to measure pressures and electrical activity (electromyography or EMG). Subjects will be asked to sit on a commode, contract (squeeze) your anal muscles, blow into a balloon, and expel the paste into the commode.

SUMMARY:
Researchers are trying to better understand why constipation occurs and improve the tests for diagnosing these conditions.

DETAILED DESCRIPTION:
Study includes a screening visit and a study day. During the initial screening visit for this study, subjects will complete three (3) questionnaires about their bowel symptoms, overall health, and anxiety and depression. A blood sample (about 4 tablespoons) will be drawn to study the relationship between genes and certain bowel habits. Subjects will be asked to provide a single stool sample to look at the bacteria in the stool.

Before the study, subjects will receive 1 to 2 Fleet's enemas to clean the rectum. After receiving the Fleet's enema (administered through a small plastic tube in the rectum), a swab attached to a small rectal catheter will be used to brush the lining of the rectum and obtain a stool specimen. Then, rectal and anal pressures will be measured by placing a small catheter (plastic tube) in the rectum, and withdrawing it slowly. Rectal sensation will be measured by inflating a small balloon in the rectum.

There are 2 procedures (rectal barostat study and fecomanoflowmetry), each of which lasts approximately 90 minutes. During the rectal barostat study, contractions will be recorded with a balloon inserted into the rectum and inflated. After the barostat study is completed, your rectum will be filled with a small amount of paste. Two thin catheters will be inserted into the anus to measure pressures and electrical activity (electromyography or EMG). Then, you will be asked to sit on a commode, contract (squeeze) your anal muscles, blow into a balloon, and expel the paste into the commode.

ELIGIBILITY:
Inclusion Criteria

* Male and female volunteers aged 18-80 years.
* Able to provide written informed consent before participating in the study.
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study.
* Individuals with chronic constipation for 1 year, with 2 or more of the following symptoms for 3 months or longer: <3 bowel motions/week, straining ≥ 25% of time, hard or lumpy stools ≥ 25% of time, anal digitation ≥ 25% of time, incomplete evacuation ≥ 25% of time, feeling of anorectal blockage ≥ 25% of time.
* Able to provide written informed consent before participating in the study.
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study.

Exclusion Criteria

* Clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns.
* Current symptoms of a functional gastrointestinal disorder assessed by questionnaire.
* Putative risk factors for pelvic floor trauma: i.e. six or more vaginal deliveries, birthweight >4500gms (macrosomia), or known 3rd or 4th degree perineal tear.
* Medications that are likely to alter gastrointestinal motility: e.g., opiates and anticholinergic medications; a stable dose of thyroxine and low doses of tricyclic agents (e.g., up to amitriptyline (50 mg daily).
* Active rectal inflammation, cancer; perianal sepsis; history of pelvic radiation, rectosigmoid surgery or inflammatory bowel disease.*
* Anxiety or depression as assessed by the Hospital Anxiety and Depression Questionnaire.
* Pregnant women, prisoners and institutionalized individuals.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-01-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rectal emptying | Baseline
  Measured by fecomanoflowmetry calculating the mean and maximum flow rate in various conditions (mg/sec), defecated volume (mg), flow time (sec) and time to maximum flow (sec). The amount of artificial stool evacuated is expressed in milligrams. The duration is in seconds. These 2 metrics are integrated to measure mg evacuated/second.
Rectoanal pressures | Baseline
  Measured by anorectal manometry in mmHg

SECONDARY OUTCOMES:
Anal sphincter electromyography (EMG) | Baseline
  Units - mV
Rectal compliance measured with a barostat | Baseline
  Pressure (mmHg) corresponding to half-maximum rectal volume during rectal distention
Rectal Capacity measured with a barostat | Baseline
  Rectal volume (ml) at maximum distending pressure during rectal distention
Rectal contractile response to distention measured with a sinusoidal oscillator | Baseline
  Rectal balloon is inflated to a preload volume of 125ml. The balloon is then oscillated around baseline volume by 25mL for 20 min at a frequency of 5 counts per minute (cpm). The mean rectal pressure (cm H2O) will be calculated over the multiple oscillation cycles within the 20 minute distention segment.
Rectal sensory threshold for first sensation to defecate using barostat balloon distention | Baseline
  The sensory threshold for first sensation to defecate is measured by stepwise inflation of the balloon (0-44 mm Hg, at 4 mm Hg increments). During this assessment participants are asked to report when they have the first sensation to defecate.
Rectal sensory threshold for desire to defecate using barostat balloon distention | Baseline
  The sensory threshold for desire to defecate is measured by stepwise inflation of the balloon (0-44 mm Hg, at 4 mm Hg increments). During this assessment participants are asked to report when they have the desire to defecate.
Rectal sensory threshold for maximum urgency during barostat balloon distention | Baseline
  The sensory threshold for maximum urgency to defecate is measured by stepwise inflation of the balloon (0-44 mm Hg, at 4 mm Hg increments). During this assessment participants are asked to report when they have the maximum urgency to defecate.
Rectal balloon expulsion time | Baseline
  During this test, the time (seconds) required to expel a water-filled rectal balloon (50 ml) will be compared between healthy people and patients

CONTACTS AND LOCATIONS:
Overall Officials: Adil E Bharucha, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials